CLINICAL TRIAL: NCT03923244
Title: Dry Eye Syndrome Description During Cataract Surgery, With Multimodal Analysis of the Ocular Surface
Acronym: C-SS0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2018 CHIAMBARETTA; 2018-A02526-49 (Other: 2018-A02526-49)
Record Dates: First submitted 2019-04-05; First posted 2019-04-22 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Dry Eye Syndrome; Ocular Surface Disease
Keywords: Dry Eye Syndrome; tear film analysis; ocular surface; cataract surgery
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Wettability

STUDY DESIGN:
Intervention Model Description: Descriptive study, interventional research involving the human person at risk and with minimal constraints (type 2), prospective, with longitudinal cohort follow-up, mono-centric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cohorte 1 (Experimental): Normal patient consultation schedule for cataract surgery with:
  * Preoperative appointment scheduled for the patient
  * Post-operative appointment 1 month before surgery No additional appointments.
  After geting consent and during the two consultations:
  * Completion of a quality of life survey by the patient. Collection of the patient's history and general and ophthalmological treatments. Questionnaire of 12 items on quality of life to be completed. For each question, the patient must answer on the frequency of the discomfort felt, from "never" to "all the time".
  * An analysis of the ocular surface is performed by a non-invasive and non-contact device for 4 minutes. This consists of taking different photographs of the eye and eyelids, allowing each to study a part of the tears.
  * Schirmer test is performed, consisting of applying the end of a small strip of blotting paper behind the lower eyelid and examining the strip after 5 minutes.
  Interventions: Diagnostic Test: OSDI survey

INTERVENTIONS:
Diagnostic Test: OSDI survey — Normal patient consultation schedule for cataract surgery with:
  * Preoperative appointment scheduled for the patient
  * Post-operative appointment 1 month before surgery No additional appointments.
  After geting consent and during the two consultations:
  * Completion of a quality of life survey by the patient. Collection of the patient's history and general and ophthalmological treatments. Questionnaire of 12 items on quality of life to be completed. For each question, the patient must answer on the frequency of the discomfort felt, from "never" to "all the time".
  * An analysis of the ocular surface is performed by a non-invasive and non-contact device for 4 minutes. This consists of taking different photographs of the eye and eyelids, allowing each to study a part of the tears.
  * Schirmer test is performed, consisting of applying the end of a small strip of blotting paper behind the lower eyelid and examining the strip after 5 minutes.
  Other Names: Schirmer test; Lacrydiag test

SUMMARY:
The main objective is to describe the characteristics of dry eye syndrome before and after surgery at one month of cataract surgery, using a multimodal analysis of the ocular surface.

The secondary objectives are to evaluate:

* Predictive factors of dry eye syndrome during cataract surgery:
* The characteristics of dry eye syndrome
* Implications for the patient's quality of life

DETAILED DESCRIPTION:
Type of study: Descriptive study, interventional research involving the human person at risk and with minimal constraints (type 2), prospective, with longitudinal cohort follow-up, mono-centric.

Number of centres: 1; The protocol will take place in the ophthalmology department of the Clermont-Ferrand University Hospital.

Study description: The study will follow the normal protocol for cataract surgery. Patients will not have any additional consultation to perform this study. The classic consultation scheme involves a preoperative appointment to set the surgical indication and inform patients about the procedure, the benefits - risks and usual follow-up.. During this consultation, the patient will have to complete a quality of life questionnaire in addition to the standard protocol, and will also have to perform a non-invasive Schirmer test and a non-contact examination of the ocular surface analysis (Lacrydiag from the Quantel laboratory, with CE marking). The patient will be seen again in a traditional post-operative consultation one month after the surgery, the same examinations will be performed.

We will use the pre and postoperative ophthalmological consultation reports, the operative report, as well as a patient questionnaire and surface analysis examination reports to conduct the study.

Main judgment criteria:

Analysis of the ocular surface defined by the study:

* OSDI questionnaire score (Ocular Surface Disease Index)
* Corneal / conjunctival states visible in slit lamp (Oxford score)
* Eyelid analysis by meibography (qualitative analysis of the eyelid glands of Meibomius and calculation of the percentage loss)
* Study of the tear film:

Lipid layer by interferometry (thickness assessment; qualitative and quantitative analysis) Aqueous layer by measuring the height of the lacrimal meniscus (quantitative analysis) Mucinic layer by evaluating the stability of the tear film (Non Invasive Break Up Time)

o Evaluation of tear secretion (Schirmer type I test)

* Eyelid analysis and tear film study will be performed simultaneously by the non-invasive test Lacrydiag.
* Definition and classification of an SSO according to different severity grades.

Secondary Judgement Criteria: Evaluate during cataract surgery:

* Predictive factors of dry eye syndrome during cataract surgery:

  * Age
  * Gender
  * General history / Systemic diseases / Eye diseases o General and topical medication use
  * Type of anesthesia used for surgery
* The characteristics of dry eye syndrome

  * Incidence of dry eye syndrome before and after surgery in our centre
  * Correlation between subjective criteria (OSDI score) and objective criteria (results of evaluation by non-invasive tests)
  * Comparison on a sample of patients (without adelphic eye pathology) in after cataract surgery between the two eyes.
* Consequences on the patient's quality of life (translated questionnaire from the Ocular Surface Disease Index from 0 to 48)

  * visual symptoms
  * activity limitations
  * adaptation to the environment
  * Post-operative satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old)
* consultants to benefit from a scheduled cataract operation at Clermont Ferrand University Hospital
* affiliation to a social security scheme
* ability to give informed consent to participate in the study.

Exclusion Criteria:

* - Patient without cataract surgery
* Congenital cataract
* Refusal to participate in the study
* Inability to answer the questionnaire (cognitive impairment, comprehension difficulties...)
* Eyelid abnormalities that may cause palpebral unocclusion
* Patient under judicial protection (guardianship, curatorship, measure to safeguard justice) or deprived of liberty
* inability to recheck the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
The main objective is to describe the characteristics of dry eye syndrome before and after surgery at one month of cataract surgery, using a multimodal analysis of the ocular surface. | Change from Baseline one month after surgery
  Definition and classification of a dry eye syndrome according to different severity grades with an analysis of the ocular surface

SECONDARY OUTCOMES:
Predictive factors of dry eye syndrome during cataract surgery | Day 1, Day 30
  Measurements with a Questionnaire to collect information about :
  * Age
  * Gender
  * General history / Systemic diseases / Eye diseases o General and topical medication
  * Type of anesthesia used for surgery
The characteristics of dry eye syndrome | Day 1, Day 30
  Incidence of dry eye syndrome before and after surgery (up to 1 month) in our centre O Correlation between subjective criteria (OSDI score) and objectives (results of evaluation by non-invasive tests)
  o Comparison on a sample of patients (without adelphic eye pathology) in cataract surgery between the two eyes to exclude any bias attributable to the measurement sequence independently of the surgery.
Consequences on the patient's quality of life (translated questionnaire from the Ocular Surface Disease Index from 0 to 48) | Day 1, Day 30
  Activity limitations
  * Adaptation to the environment
  * Post-operative satisfaction at one month For each question, the patient must answer on the frequency of the discomfort felt, from "never" to "all the time". After calculation, a score between 0 and 100 is obtained. Consensually, it is considered that the drought syndrome is obvious when the score is 18 or more, and that it is a severe from 33 to 35.

CONTACTS AND LOCATIONS:
Overall Officials: frédéric Chiambaretta, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France